CLINICAL TRIAL: NCT02288962
Title: Dopamine Agonist Treatment of Non-functioning Pituitary Adenomas (NFPAs) - a Randomized Controlled Trial
Brief Title: Dopamine Agonist Treatment of Non-functioning Pituitary Adenomas
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012/677; 2012-001338-32 (EudraCT Number)
Record Dates: First submitted 2014-11-05; First posted 2014-11-13 (Estimated); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Pituitary Neoplasms; Adenoma
Keywords: dopamine agonists; cabergoline
MeSH Terms: conditions — Pituitary Neoplasms; Adenoma | interventions — Cabergoline

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cabergoline (Experimental): Target dose for cabergoline is 2 mg/week.The medication is administered in the evening to minimize side effects. If intolerable side effects occur despite this, it may be necessary to treat with a lower dose than 2 mg per week.
  Treatment scheme: 0.5 mg x 1 per week the first 2 weeks, then 0.5 mg x 2 per week the next 2 weeks, then 1 + 0.5 mg per week the next 2 weeks, then 1 mg x 2 per week (target dose) for the rest of the study
  Interventions: Drug: cabergoline
- observation (No Intervention): visits and controls as usual

INTERVENTIONS:
Drug: cabergoline
  Other Names: galastop; FCE 21336; Cabaser; Dostinex; Cabaseril; cabergoline diphosphate
  Arms: cabergoline

SUMMARY:
Due to lack of hormone overproduction in non-functioning pituitary adenomas (NFPAs), only the symptomatic adenomas or large adenomas with proven growth and risk for symptoms in near future will undergo pituitary surgery. The remaining adenomas are monitored regularly. Operation of these large adenomas will rarely remove all tumour tissue, and there is also a risk of worsening of pituitary function. Often, adenomas with the highest growth potential are operated several times and some also need radiation therapy, providing additional risk for pituitary failure. Unlike some of the hormone-producing adenomas, there is no established pharmacological treatment for NFPAs. However, there are a few non-randomized studies suggesting that treatment with dopamine agonists may slow growth, and also induce tumour shrinkage. At present, cabergoline is the dopamine agonist most widely used in the treatment of pituitary adenomas secreting prolactin.

Aim is to study the effect of medical treatment with cabergoline in non-functioning pituitary adenomas on the change in tumour volume.

ELIGIBILITY:
Inclusion Criteria:

* A previously untreated non-functioning pituitary macroadenoma (largest diameter ≥ 10 mm) with either demonstrated growth on repeated MRI scans or ≤ 2 mm distance to chiasma opticum, or:
* a residual non-functioning pituitary adenoma after surgery (largest diameter ≥ 5 mm) that is either extrasellar and/or with documented growth after surgical treatment of a non-functioning pituitary macroadenoma

Exclusion Criteria:

* Clear indication for surgery at the time of inclusion
* Previous radiation therapy
* Pituitary surgery the last 6 months
* Previous apoplexy/bleeding in the adenoma
* Pregnancy or lactation
* Contraindications for cabergoline treatment (Known cardiac valvular disease, known pulmonal, pericardial or retroperitoneal fibrosis, clinical significant liver insufficiency, use of medications that interact with cabergoline
* unfit to participate due to any other reason

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
change in tumour volume during the main study of two years | 2 years
  This includes the percentage and absolute change in tumour volume, but also the number of patients with significant tumour shrinkage or tumour growth (defined by ≥ 10 % or ≥ 2 mm shrinkage/growth in at least one dimension)

SECONDARY OUTCOMES:
need for surgical and/or radiation treatment | up till 2 years
changed pituitary function | up till 2 years
  measured by analysis of blood tests, basal and stimulation tests
change in tumour's distance to chiasma opticum in mm | up till 2 years
  as measured by analysis of MRI images
development of cardiac valvulopathy | up till 2 years
  as measured by analysis of echo cardiography
impulse control disorder | up till 2 years
  as measured by questionnaire visual files: clinical evaluation by ophthalmologist and perimetry

CONTACTS AND LOCATIONS:
Overall Officials: Sven M Carlsen, prof md, Principal Investigator — Norwegian University of Science and Technology
Locations (3):
- Norway (2):
  - Department of Endocrinology, Akershus University hospital, Oslo
  - Department of Endocrinology, St. Olavs Hospital, Trondheim
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No